CLINICAL TRIAL: NCT00093743
Title: Low-Dose Total Body Irradiation and Fludarabine Followed By Unrelated Donor Stem Cell Transplantation for Patients With Fanconi Anemia - A Multicenter Trial
Brief Title: Low-Dose Total-Body Irradiation and Fludarabine Phosphate Followed by Unrelated Donor Stem Cell Transplant in Treating Patients With Fanconi Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1444.00; NCI-2012-00593 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1444.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Childhood Acute Myeloid Leukemia in Remission; Childhood Myelodysplastic Syndromes; Fanconi Anemia; Previously Treated Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities; Fanconi Anemia | interventions — fludarabine phosphate; Cyclosporine; Whole-Body Irradiation; Transplantation; Peripheral Blood Stem Cell Transplantation; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (allogeneic bone marrow or PBSC transplantation) (Experimental): NON-MYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2, cyclosporine IV every 8-12 hours on days -3 to 0, and undergo low-dose TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic bone marrow or PBSC transplantation on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO or IV every 8-12 hours on days 1-100 with taper to day 177, and mycophenolate mofetil PO or IV every 8 hours on days 0-40 with taper to day 96.
  Interventions: Drug: fludarabine phosphate; Drug: cyclosporine; Radiation: total-body irradiation; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic bone marrow transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSC transplantation
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBSC transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: mycophenolate mofetil — Given PO or IV
  Other Names: Cellcept; MMF

SUMMARY:
Based on success in other diseases, the Fred Hutchinson Cancer Research Center (FHCRC) has developed a transplant procedure for Fanconi anemia (FA), which does not completely destroy the patient's remaining bone marrow. It should also be less harmful (toxic). Researchers wish to test whether this approach can overcome the graft failure often seen when bone marrow or peripheral blood stem cells from an unrelated donor are used. Researchers also will look at whether the procedure is less toxic than a conventional bone marrow transplant (BMT).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether donor chimerism can be achieved in patients with Fanconi anemia receiving marrow or peripheral blood stem cell (PBSC) grafts from unrelated donors following low dose total body irradiation (TBI), fludarabine (fludarabine phosphate), mycophenolate mofetil, and cyclosporine.

II. To determine the lowest dose of TBI necessary to achieve donor chimerism in at least 80% of patients.

III. To determine the incidence of severe regimen-related toxicity.

SECONDARY OBJECTIVES:

I. To determine the survival of Fanconi anemia patients transplanted with unrelated donor marrow or PBSC grafts after conditioning with a non-myeloablative regimen.

II. To determine the incidence and severity of graft-vs-host disease (GVHD) incurred with unrelated bone marrow or PBSC grafts transplant patients with Fanconi anemia.

III. To determine if mixed chimerism results in amelioration of symptoms associated with bone marrow failure in patients with Fanconi anemia.

OUTLINE:

NON-MYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -4 to -2, cyclosporine IV every 8-12 hours on days -3 to 0, and undergo low-dose TBI on day 0.

TRANSPLANTATION: Patients undergo allogeneic bone marrow or PBSC transplantation on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) or IV every 8-12 hours on days 1-100 with taper to day 177, and mycophenolate mofetil PO or IV every 8 hours on days 0-40 with taper to day 96.

After completion of study treatment, patients are followed up at 6 months and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with marrow failure and increased chromosome fragility as determined in the diepoxybutane (DEB) or mitomycin C test
* Any patient with Fanconi anemia (FA) with marrow failure meeting the following criteria:
* Granulocyte count < 0.2 x 10^9/L
* Platelet count < 20 x 10^9/L
* Hemoglobin < 8 g/dl
* Corrected reticulocyte count <1%
* Any patient with FA as determined by DEB fragility, who has life-threatening marrow failure involving a single hematopoietic lineage
* Any patient with FA and pre-existing cytogenetic abnormality including hematopoietic malignancy (myelodysplastic syndromes [MDS] or acute myeloid leukemia [AML]) in remission
* DONOR: Unrelated Donors who are prospectively: Matched for human lymphocyte antigen (HLA)-DRB1 and DQB1 alleles (must be defined by high resolution typing); only a single allele disparity will be allowed for HLA -A, B, or C as defined by high resolution typing
* DONOR: HLA typing will be performed at the highest level of resolution available at the time of transplant

Exclusion Criteria:

* Evidence for hematopoietic malignancy in relapse
* Heart or lung disease that would prevent compliance with conditioning and GvHD regimen or would severely limit the probability of survival
* Human immunodeficiency virus (HIV) seropositive patients
* Females who are pregnant or breastfeeding, or unwilling to use contraceptive techniques during and for the 12 months following treatment
* DONOR: Donors who by DEB testing are found to have FA
* DONOR: Donors who test positive in the lymphocytotoxic crossmatch assay
* DONOR: Donors who are HIV positive
* DONOR: Donors who for other medical or psychological reasons are not suitable as donors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2000-01; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Engraftment, defined as donor chimerism (mixed or complete) | Day 28
  Mixed chimerism is defined as presence of 5-95%, complete chimerism as > 95% donor derived cells in the peripheral blood. Patient data will be summarized using standard statistical methods.
Engraftment, defined as donor chimerism (mixed or complete) | Day 56
  Mixed chimerism is defined as presence of 5-95%, complete chimerism as > 95% donor derived cells in the peripheral blood. Patient data will be summarized using standard statistical methods.
Engraftment, defined as donor chimerism (mixed or complete) | Day 84
  Mixed chimerism is defined as presence of 5-95%, complete chimerism as > 95% donor derived cells in the peripheral blood. Patient data will be summarized using standard statistical methods.
Engraftment, defined as donor chimerism (mixed or complete) | Day 180
  Mixed chimerism is defined as presence of 5-95%, complete chimerism as > 95% donor derived cells in the peripheral blood. Patient data will be summarized using standard statistical methods.
Regimen toxicity assessed using the Bearman scale | Up to day 100
  Patient data will be summarized using standard statistical methods.
Acute GvHD defined using the Seattle criteria | Day 84
  For the evaluation of GvHD, time of onset, severity, and treatment will be recorded. Patient data will be summarized using standard statistical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Kiem, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (5):
- United States (5):
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington